CLINICAL TRIAL: NCT00968006
Title: Effects of 4-week Sitagliptin Therapy on Endothelial Progenitor Cells in Type 2 Diabetic Patients. A Non-randomized Controlled Open-label Pilot Trial.
Brief Title: Effect of Sitagliptin on Endothelial Progenitor Cells
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Padova (Other)
Responsible Party: Angelo Avogaro, Associate Professor (PI), Dept Clinical and Experimental Medicine, University of Padova Medical School
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: Sita-EPC
Record Dates: First submitted 2009-08-26; First posted 2009-08-28 (Estimated); Last update posted 2010-04-05 (Estimated); Status verified 2010-04

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: diabetes; endothelium; stem cells
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): Sitagliptin 100 mg once daily for 4 weeks
  Interventions: Drug: Sitagliptin
- Control (No Intervention): No change in anti-diabetic treatment regimen for at least 4 weeks.

INTERVENTIONS:
Drug: Sitagliptin — 100 mg once daily for 4 weeks
  Other Names: Januvia; Xelevia; Tesavel
  Arms: Treatment

SUMMARY:
Endothelial progenitor cells (EPCs) are involved in cardiovascular homeostasis, through angiogenesis and endothelial healing. Diabetic patients have a high risk of cardiovascular events and low levels of circulating EPCs.

Sitagliptin is an oral DPP-IV antagonist, approved for the treatment of type 2 diabetes. It increases the bioavailability of endogenous incretins, thus improving insulin and glucagon secretion. SDF-1, one of the major EPC regulators, is also a substrate of DPP-IV. This study tests the hypothesis that sitagliptin increases the levels of circulating EPCs in type 2 diabetic patients.

DETAILED DESCRIPTION:
Diabetic patients suffer an elevated wirk of cardiovascular events, which strongly impact on morbidity and mortality. The mechanisms that lead to cardiovascular disease in diabetes include alterations in the endothelial layer, due to hyperglycemia, oxidative stress and other associated abnormalities. Endothelial progenitor cells (EPCs) are bone marrow-derived cells involved in endothelial repair after injury, and they have been found to be reduced in diabetic patients. Thus, reduced EPCs in diabetes may be another mechanism of vascular disease induction. Reduction of EPCs in diabetes is attributable at least in part to the impairment of bone marrow mobilization, which is regulated by the chemokine SDF-1alpha, among others.

The oral hypoglycemia agent sitagliptin is a dipeptidyl dipeptidase-IV inhibitor, which prevents degradation of endogenous incretins (GIP and GLP-1), thus re-equilibrating insulin and glucagon secretion. Sitagliptin may also increase the concentrations of SDF-1alpha, which is another substrate of DPP-IV. The hypothesis is that sitagliptin may increase circulating EPC levels, through SDF-alpha.

This is going to be a pilot, non-randomized controlled 4-week trial of 100 mg oral sitagliptin therapy added to metformin/sulphonylureas in poorly controlled type 2 diabetic patients. At baseline and 4 weeks after the initiation of therapy blood samples will be drawn for the determination of circulating EPC levels, and concentrations of SDF-1alpha. EPCs will be defined as CD34+KDR+ cells and measured by flow cytometry as previously described in detail. SDF-1alpha will be measured using ELISA kits according to the manufacturer's instructions.

Changes between baseline and 4 weeks will be evaluated using two-tailed paired Student's t test and statistical significance accepted at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes;
* Both genders
* Age 40-80
* fasting c-peptide >=1.0 ng/L
* Therapy with metformin or sulphonylureas
* HbA1c >7.0%
* No contraindications to sitagliptin use

Exclusion Criteria:

* Type 1 diabetes
* Age <40 or >80
* fasting c-peptide <1.0 ng/L
* Therapy with TZD
* HbA1c <=7.0%
* Acute concomitant diseases
* Immunological disorders
* Recent (within 3 months) cardiovascular events or surgery
* Pregnancy and lactation
* Inability to provide informed consent

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Change in circulating CD34+KDR+ endothelial progenitor cells | 4 weeks

SECONDARY OUTCOMES:
Change in SDF-1alpha concentrations | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Avogaro, MD PhD, Principal Investigator — Dept. Clinical and Experimental Medicine, University of Padova, Medical School, Padova (Italy)
Locations (1):
- University of Padova, Medical School, Padua, Italy

REFERENCES:
- [Result] Fadini GP, Boscaro E, Albiero M, Menegazzo L, Frison V, de Kreutzenberg S, Agostini C, Tiengo A, Avogaro A. The oral dipeptidyl peptidase-4 inhibitor sitagliptin increases circulating endothelial progenitor cells in patients with type 2 diabetes: possible role of stromal-derived factor-1alpha. Diabetes Care. 2010 Jul;33(7):1607-9. doi: 10.2337/dc10-0187. Epub 2010 Mar 31. PMID 20357375